CLINICAL TRIAL: NCT06883383
Title: Data Analysis and Evaluation of the Incidence of Life-threatening Ventricular Arrhythmias in Patients with Newly Diagnosed Cardiomyopathies of NICM or MI/CAD Origin PROTECTED from SCD by a WCD
Acronym: SCD-PROTECT
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Zoll CMS GmbH (Unknown)
Responsible Party: Principal Investigator, David Duncker, Head of Hannover Heart Rhythm Center, Department of Cardiology and Angiology, Hannover Medical School
Other Study IDs: SCD-PROTECT
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cardiomyopathy (Ischemic or Non-Ischemic)
Keywords: sudden cardiac arrest; sudden cardiac death; non-ischemic cardiomyopathy; dilated cardiomyopathy; wearable cardioverter-defibrillator; left ventricular ejection fraction; ischemic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Ischemia; Death, Sudden, Cardiac; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
SCD-PROTECT is an epidemiological, observational, multicenter study to assess the incidence of sudden cardiac arrest/death (SCA/SCD) in patients with newly diagnosed non-ischemic cardiomyopathy or with myocardial infarction/coronary artery disease. Data on SCA/SCD risk in the early phase of disease, especially during medication up-titration while left ventricular ejection fraction is reduced, are sparse.

DETAILED DESCRIPTION:
SCD-PROTECT is an epidemiological, observational, multicenter study, evaluating the incidence of sudden cardiac arrest (SCA) / sudden cardiac death (SCD) in patients with reduced left ventricular ejection fraction (LVEF) due to newly diagnosed non-ischemic cardiomyopathy (NICM) or a myocardial infarction/coronary artery disease with intervention (MI/CAD). In the early phase (3 months) during up-titration of guideline-recommended therapy (GRMT) a wearable cardioverter defibrillator (WCD) can be indicated due to increased risk for SCA/SCD in these patients. The WCD provides continuous arrhythmia monitoring, detection of life-threatening ventricular arrhythmias, and provides automatic defibrillation within a minute of detection of a potentially fatal ventricular tachyarrhythmia whatever the cause of increased risk of SCD. Currently, detailed data for risk of SCA/SCD in patients with NICM or MI/CAD during the early phase are sparse.

The SCD-PROTECT study is a comprehensive, nationwide analysis of at least 18.000 consecutive patients using a WCD (LifeVest®, ZOLL, Pittsburgh, PA, USA) in Germany to evaluate the risk of SCA/SCD in the early phase of disease.

All patients who received a WCD (LifeVest®, ZOLL, Pittsburgh, PA, USA) from December 2021 to May 2023 in Germany will be screened for inclusion. Observation period will start with first ECG recording of the WCD and terminates with individual end-of-WCD-use. Primary objective is the SCA/SCD incidence, measured by the percentage of patients with at least one appropriate treatment (appropriate shock) delivered and automatically recorded by WCD. The incidence density of appropriate shocks per 100 patient years will also be calculated.

Secondary objectives include inappropriate WCD treatments, mortality and side effects during WCD wearing time. Exploratory objectives are trajectory of LVEF, compliance with WCD use, time to first appropriate shock from beginning of wearing time until first WCD shock and incidences of appropriate shocks (primary endpoint) by subtype of NICM or MI/CAD.

NICM and MI/CAD sub-types are categorized by the investigator team at baseline and may include the following: DCM, Myocarditis, PPCM, Tako-Tsubo CM, Tachymyopathy, Toxic CM, Sarcoidosis Genetic/Congenital, and others vs. Post Myocardial Infarction, Coronary Heart Disease and others.

Patient data are extracted from routinely collected medical records by analysts, blinded to the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older.
* Subjects must be prescribed a WCD for a high risk of SCD.
* Subjects must have been fitted with a WCD, and a baseline for ECG-analysis must have been established.
* Subjects must have worn the WCD; time zero of inclusion is the activation of the ECG.
* Subjects must have had a diagnosis of newly diagnosed NICM or MI/CAD with reduced LVEF as indication for WCD prescription.

Exclusion Criteria:

* No specific exclusion criteria will be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes consecutively all patients with NICM or MI/CAD diagnosis and WCD usage (LifeVest®, ZOLL, Pittsburgh, PA, USA) in Germany. The Zoll database systematically registers all patients who are prescribed the LifeVest® in Germany. For this study, data from the ZPM (Zoll Patient Management System), which holds the recordings of the WCD is also integrated to assess treatments and compliance.
  All patients with NICM or MI/CAD indication, entered in the ZOLL database since December 2021 will be enrolled retrospectively into the study. From January 2023 to May 2023 patients will be prospectively enrolled following the same protocol.
Sampling Method: Probability Sample
Enrollment: 19598 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of SCD/SCA | Observation period starts with baseline of WCD-use and continues through end of WCD-use, an average of 2-3 months
  Incidence of patients with NICM or MI/CAD with at least one appropriate treatment (appropriate shock) observed during WCD-use. Treatment events will be automatically recorded through the monitoring device. The incidence density of appropriate shocks per 100 patient years will also be calculated.

SECONDARY OUTCOMES:
Incidence of inappropriate shocks | Observation period starts with baseline of WCD-use and continues through end of WCD-use, an average of 2-3 months
  Percentage of patients with inappropriate shocks observed during WCD-use. Events will be automatically recorded through the monitoring device.
Mortality | Observation period starts with baseline of WCD-use and continues through end of WCD-use, an average of 2-3 months
  Percentage of death during observation period
Adverse events | Observation period starts with baseline of WCD-use and continues through end of WCD-use, an average of 2-3 months
  Adverse events during observation period

OTHER OUTCOMES:
Average WCD wear-time in days | Observation period starts with baseline of WCD-use and continues through end of WCD-use, an average of 2-3 months
  Average WCD wear-time in days, from baseline until end of WCD-use, measured in days
WCD compliance | Observation period starts with baseline of WCD-use and continues through end of WCD-use, an average of 2-3 months
  Compliance, meaning average wear-time of the WCD per day, measured in hours per day.
Cumulative Incidences of appropriate treatments per sub-etiologies | Observation period starts with baseline of WCD-use and continues through end of WCD-use, an average of 2-3 months
  Cumulative Incidences of appropriate treatments per sub-etiologies, measured in events per 100 patient-years
Time from baseline of WCD-use until first appropriate WCD-treatment | From baseline of WCD-use until first appropriate treatment by the WCD, assessed through end of WCD use, an average of 2-3 months
  Time from baseline of WCD-use until first appropriate WCD-treatment, measured in days
Trajectory of left ventricular ejection fraction (LVEF) | Pre-hospital (up to one year), at hospital discharge (assessed up to 3 days), and at end of WCD use (an average of 2-3 months from base line)
  Trajectory of left ventricular ejection fraction (LVEF), measured in percent LVEF at the time-points pre-hospital, at hospital discharge (corresponding to baseline of WCD-use), and at end of WCD-use

CONTACTS AND LOCATIONS:
Overall Officials: Johann Bauersachs, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No